CLINICAL TRIAL: NCT04313712
Title: A Pre-post Study Evaluating the Safety and Efficacy of Ibogaine-Magnesium Therapy in Veterans With Sequelae of Repeated Blast Exposure
Brief Title: Pre-post Evaluation of the Safety and Efficacy of Ibogaine-Magnesium Therapy in Veterans With Repeated Blast Exposure
Status: Active, not recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Nolan R, Assistant Professor, Stanford University, Stanford University
Other Study IDs: 54095
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Blast or Combat Exposure; Head Injury Trauma
Keywords: blast exposure; combat exposure; head trauma
MeSH Terms: conditions — Craniocerebral Trauma | interventions — Ibogaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: All study participants will be observed before and after they receive ibogaine-magnesium therapy.
  Interventions: Drug: ibogaine with magnesium treatment

INTERVENTIONS:
Drug: ibogaine with magnesium treatment — Participants will receive magnesium sulfate intravenously and ibogaine orally.

SUMMARY:
A Pre-post Study Evaluating the Safety and Efficacy of Ibogaine-Magnesium Therapy in Veterans with Sequelae of Repeated Blast Exposure.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a leading cause of disability worldwide and is particularly common among combat veterans. Deleterious sequelae can include functional impairments and comorbid psychiatric syndromes such as posttraumatic stress disorder (PTSD), depression, and anxiety. Special Operations Forces Veterans (SOV) may be at an elevated risk for these complications, leading some to seek treatment alternatives like the oneirogen ibogaine despite limited evidence of safety or efficacy.

We will assess the safety profile of the compound by assessing unexpected or serious adverse events.

The primary outcome will be change in the World Health Organization Disability Assessment Schedule 2.0 (WHODAS) from baseline to post-treatment, with change from baseline to the one-month follow-up a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female veteran, 18 to 70 years of age, inclusive, at screen.
2. Able to read, understand, and provide written, dated informed consent prior to screening. Participants will be deemed likely to comply with the study protocol and communicate with study personnel about adverse events and other clinically important information.
3. Has a history of head trauma, combat or blast exposure.
4. Scheduled themselves for ibogaine-magnesium therapy at Nouvelle Vie in Mexico.
5. Participants must be willing and able to travel to Stanford University before and after ibogaine-magnesium therapy.
6. Capable of getting an MRI scan.
7. Willing to be video recorded during the consenting process. (to be stored on a secure server, no PHI associated with video recordings)
8. Body mass index between 17-35kg/m2.
9. If female, a status of non-childbearing potential or use of an acceptable form of birth control per the following specific criteria:

   1. Non-childbearing potential (e.g., physiologically incapable of becoming pregnant, i.e., permanently sterilized (status post hysterectomy, bilateral tubal ligation), or is post-menopausal with her last menses at least one year prior to screening); or
   2. Childbearing potential, and meets the following criteria:

   i. Childbearing potential, including women using any form of hormonal birth control, on hormone replacement therapy started prior to 12 months of amenorrhea, using an intrauterine device (IUD), having a monogamous relationship with a partner who has had a vasectomy, or is sexually abstinent.

   ii. Negative urinary pregnancy test at screening, confirmed by a negative urinary pregnancy test at randomization prior to receiving study treatment.

   iii. Willing and able to continuously use one of the following methods of birth control during the course of the study, defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly: implants, injectable or patch hormonal contraception, oral contraceptives, IUD, double-barrier contraception, sexual abstinence. The form of birth control will be documented at screening and baseline.
10. Participants must be US citizens.

Exclusion Criteria:

1. Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study.
2. Female that is pregnant or breastfeeding.
3. Claustrophobic.
4. History of a neurological disorder (i.e. Parkinson's, epilepsy, dementia, etc.) excluding sequelae of traumatic injury.
5. In the judgment of the investigator, the subject is at significant risk for suicidal behavior during the course of their participation in the study.
6. History of schizophrenia or schizoaffective disorders, or any history of psychotic symptoms.
7. Has a clinically significant abnormality on the screening physical examination that might affect safety, study participation, or confound interpretation of study results.
8. Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation.
9. Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation.
10. Any history of cardiovascular problems.
11. Any history of liver or kidney problems.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans with a history of head trauma, combat or blast exposure that have arranged for ibogaine-magnesium therapy in other countries.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change in score on the WHODAS 2.0 | Baseline to immediate post visit.
  The WHODAS 2.0 is a generic assessment of disability across six domains of functioning including cognition, mobility, self-care, interpersonal relationships, life activities, and community activities. The higher the score, the greater the level of self-reported disability in functioning. Scores from baseline will be compared to scores at the immediate post-treatment.

SECONDARY OUTCOMES:
Change in score on the WHODAS 2.0 | Baseline to 1-month post visit.
  The WHODAS 2.0 is a generic assessment of disability across six domains of functioning including cognition, mobility, self-care, interpersonal relationships, life activities, and community activities. The higher the score, the greater the level of self-reported disability in functioning. Scores from baseline will be compared to scores at 1-month post-visit.

CONTACTS AND LOCATIONS:
Overall Officials: Nolan Williams, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Cherian KN, Keynan JN, Anker L, Faerman A, Brown RE, Shamma A, Keynan O, Coetzee JP, Batail JM, Phillips A, Bassano NJ, Sahlem GL, Inzunza J, Millar T, Dickinson J, Rolle CE, Keller J, Adamson M, Kratter IH, Williams NR. Magnesium-ibogaine therapy in veterans with traumatic brain injuries. Nat Med. 2024 Feb;30(2):373-381. doi: 10.1038/s41591-023-02705-w. Epub 2024 Jan 5. PMID 38182784